CLINICAL TRIAL: NCT05358158
Title: Efficacy of Avoiding Chest Drain After Video-assisted Thoracoscopic Surgery Wedge Resection
Brief Title: Chest dRain rEmoval intrAoperatively afTer thoracOscopic Wedge Resection
Acronym: CREATOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Lin Huang, Department of cardiothoracic surgery, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21012837
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Lung Neoplasms; Lung Surgery; Enhanced Recovery After Surgery; Fast-track Surgery; Pain; Opioid Use; Remission
MeSH Terms: conditions — Lung Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain-free group (Experimental): Participants undergoing video-assisted thoracoscopic wedge resection with a positive intraoperative sealing test are treated with intraoperative chest tube removal.
  Interventions: Procedure: Intraoperative air leak test; Procedure: Intraoperative chest drain removal
- Chest drain group (Active Comparator): Participants undergoing video-assisted thoracoscopic wedge resection with a positive intraoperative sealing test are treated with a standard postoperative chest tube.
  Interventions: Procedure: Intraoperative air leak test; Procedure: Standard chest drain placement

INTERVENTIONS:
Procedure: Intraoperative air leak test — A standard 28 Fr chest drain is inserted through the anterior port hole with all port holes closed. With the tip of the chest tube below water, the pleura is emptied from air during continuous ventilation of the lungs. An air leak after 5 minutes of ventilation indicates a negative sealing test, whereas a cessation of air leak within 5 minutes indicates a positive sealing test.
Procedure: Intraoperative chest drain removal — Chest drain is removed intraoperatively.
  Arms: Drain-free group
Procedure: Standard chest drain placement — Chest drain is left in pleura.
  Arms: Chest drain group

SUMMARY:
Chest drain is used routinely after lung surgery. Despite preliminary studies demonstrate the feasibility and safety of intraoperative chest drain removal, these are either retrospective or mainly concerning benign disease.

Hypothesis: Participants treated without post-operative chest tube after thoracoscopic wedge resection have less pain, reduced opioid usage without increasing postoperative complications than participants treated with standard post-operative chest tube, and could possibly be discharged earlier.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients referred for elective three port video-assisted thoracoscopic surgery wedge resection of the lung for suspected or confirmed malignant nodules.
* first second forced expiratory volume ≥60% of expected.
* No increased bleeding risk (e.g. preoperative international normalized ratio >2, overdue discontinuation of anticoagulants according to guidelines by the Danish Society for Thrombosis and Haemostasis, known coagulopathy).
* Not scheduled for frozen section pathology of wedge resection and subsequent lobectomy.
* Able and willing to give informed consent.

Exclusion Criteria:

* Increased risk of post-operative air leak assessed perioperatively by the surgeon (e.g. severe adhesions, bullous/emphysematous lung tissue, defects of the visceral pleura due to iatrogenic or other reasons, suturing in the lung tissue, deep lung resection).
* Increased risk of post-operative bleeding assessed perioperatively by the surgeon (e.g. intraoperative bleeding or oozing).
* Air leak during intraoperative air leak test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-03-17 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Acute Pain | Up to postoperative day 1
  Postoperative pain assessed in three different situations (at rest, arms lifted and during cough) by questionnaire at 3 and 6 hours after surgery, and on the morning of postoperative day 1 at 8 a.m
Rescue analgesics | Up to postoperative day 1
  The amount of rescue analgesics given assessed as cumulative amount of morphine during the first 24 hours after surgery milligram equivalents (MME) as defined by pro.medicine.dk hosted by the Danish Association of the Pharmaceutical Industry

SECONDARY OUTCOMES:
Pneumothorax | Up to postoperative 2 weeks
  Number and size of pneumothorax at 6 hours after surgery in the drain-free group, 2 hours after drain removal in the drain group, and postoperative 2-week for both
Complications | Up to postoperative day 30
  Surgical and medical complications including mortality
Chest drain reinsertion | Up to postoperative day 30
  Number and reasons of chest drain reinsertion
Length of stay | Through post-operative discharge, an average of 2 days
  Days in hospital after index surgery
Time to fulfilled discharge criteria | Through post-operative discharge, an average of 2 days
  Days to meet discharge criteria but stay in hospital
Readmission | Through post-operative admission, an average of 7 days
  Number and reasons of readmissions
Quality of recovery after surgery | Up to postoperative day 1
  Evaluate patients' quality of life by questionnaire before surgery, at the first day after surgery
Standard analgesics given | Up to postoperative 2 weeks
  Number of patients who did not receive planned postoperative analgesics according to the standards at their institution
Persistent pain | Up to postoperative day 6
  Postoperative pain assessed in three different situations (at rest, arms lifted and during cough) by questionnaire from postoperative day 2 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: René H Petersen, MD, PhD, Study Chair — Rigshospitalet, Denmark; Thomas D Christensen, MD, PhD, Study Director — Aarhus University Hospital; Bo L Holbek, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Morten Bendixen, MD, PhD, Principal Investigator — Aarhus University Hospital; Jonas J Rasmussen, MD, Principal Investigator — Aarhus University Hospital; Henrik Kehlet, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Henrik J Hansen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Thomas Decker Christensen, Aarhus, Aarhus N
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication are planned to share to other researchers if they connect with the corresponding author of the publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The time when summary data are published.
Access Criteria: Others who need the IPD and relevant information should ask the correspoding author of the publication

REFERENCES:
- [Result] Cerfolio RJ, Bryant AS. The management of chest tubes after pulmonary resection. Thorac Surg Clin. 2010 Aug;20(3):399-405. doi: 10.1016/j.thorsurg.2010.04.001. PMID 20619231
- [Result] Luckraz H, Rammohan KS, Phillips M, Abel R, Karthikeyan S, Kulatilake NE, O'Keefe PA. Is an intercostal chest drain necessary after video-assisted thoracoscopic (VATS) lung biopsy? Ann Thorac Surg. 2007 Jul;84(1):237-9. doi: 10.1016/j.athoracsur.2007.03.007. PMID 17588421
- [Result] Holbek BL, Horsleben Petersen R, Kehlet H, Hansen HJ. Fast-track video-assisted thoracoscopic surgery: future challenges. Scand Cardiovasc J. 2016;50(2):78-82. doi: 10.3109/14017431.2015.1114665. Epub 2015 Dec 1. PMID 26514281
- [Result] Refai M, Brunelli A, Salati M, Xiume F, Pompili C, Sabbatini A. The impact of chest tube removal on pain and pulmonary function after pulmonary resection. Eur J Cardiothorac Surg. 2012 Apr;41(4):820-2; discussion 823. doi: 10.1093/ejcts/ezr126. Epub 2011 Dec 21. PMID 22219425
- [Result] Mao M, Hughes R, Papadimos TJ, Stawicki SP. Complications of chest tubes: a focused clinical synopsis. Curr Opin Pulm Med. 2015 Jul;21(4):376-86. doi: 10.1097/MCP.0000000000000169. PMID 26016583
- [Result] Bardell T, Petsikas D. What keeps postpulmonary resection patients in hospital? Can Respir J. 2003 Mar;10(2):86-9. doi: 10.1155/2003/610570. PMID 12693389
- [Result] Wildgaard K, Petersen RH, Hansen HJ, Moller-Sorensen H, Ringsted TK, Kehlet H. Multimodal analgesic treatment in video-assisted thoracic surgery lobectomy using an intraoperative intercostal catheter. Eur J Cardiothorac Surg. 2012 May;41(5):1072-7. doi: 10.1093/ejcts/ezr151. Epub 2011 Dec 21. PMID 22219442
- [Result] Watanabe A, Watanabe T, Ohsawa H, Mawatari T, Ichimiya Y, Takahashi N, Sato H, Abe T. Avoiding chest tube placement after video-assisted thoracoscopic wedge resection of the lung. Eur J Cardiothorac Surg. 2004 May;25(5):872-6. doi: 10.1016/j.ejcts.2004.01.041. PMID 15082297
- [Result] Koc T, Routledge T, Chambers A, Scarci M. Do patients undergoing lung biopsy need a postoperative chest drain at all? Interact Cardiovasc Thorac Surg. 2010 Jun;10(6):1022-5. doi: 10.1510/icvts.2010.232892. Epub 2010 Mar 22. PMID 20308263
- [Result] Holbek BL, Hansen HJ, Kehlet H, Petersen RH. Thoracoscopic pulmonary wedge resection without post-operative chest drain: an observational study. Gen Thorac Cardiovasc Surg. 2016 Oct;64(10):612-7. doi: 10.1007/s11748-016-0692-6. Epub 2016 Aug 10. PMID 27510705
- [Result] Park JB, Hwang JJ, Lee WS, Kim YH, Lee SA. Postoperative chest tube placement after thoracoscopic wedge resection of lung for primary spontaneous pneumothorax: is it mandatory? J Thorac Dis. 2018 Aug;10(8):4812-4818. doi: 10.21037/jtd.2018.07.13. PMID 30233854
- [Result] Liao HC, Yang SM, Hung MH, Cheng YJ, Hsu HH, Chen JS. Thoracoscopic Surgery Without Drainage Tube Placement for Peripheral Lung Nodules. Ann Thorac Surg. 2020 Mar;109(3):887-893. doi: 10.1016/j.athoracsur.2019.10.048. Epub 2019 Dec 13. PMID 31843633
- [Result] Lesser T, Doenst T, Lehmann T, Mukdessi J. Lung Bioposy Without Pleural Drainage. Dtsch Arztebl Int. 2019 May 10;116(19):329-334. doi: 10.3238/arztebl.2019.0329. PMID 31288906
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. Trials. 2010 Mar 24;11:32. doi: 10.1186/1745-6215-11-32. PMID 20334632
- [Result] Altman DG, Bland JM. Statistics notes: the normal distribution. BMJ. 1995 Feb 4;310(6975):298. doi: 10.1136/bmj.310.6975.298. No abstract available. PMID 7866172
- [Result] Bland JM, Altman DG. The use of transformation when comparing two means. BMJ. 1996 May 4;312(7039):1153. doi: 10.1136/bmj.312.7039.1153. No abstract available. PMID 8620137
- [Result] Hickey GL, Dunning J, Seifert B, Sodeck G, Carr MJ, Burger HU, Beyersdorf F; EJCTS and ICVTS Editorial Committees. Statistical and data reporting guidelines for the European Journal of Cardio-Thoracic Surgery and the Interactive CardioVascular and Thoracic Surgery. Eur J Cardiothorac Surg. 2015 Aug;48(2):180-93. doi: 10.1093/ejcts/ezv168. Epub 2015 May 12. PMID 25971435
- [Result] Bland JM, Altman DG. Correlation, regression, and repeated data. BMJ. 1994 Apr 2;308(6933):896. doi: 10.1136/bmj.308.6933.896. No abstract available. PMID 8173371
- [Result] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Kleif J, Edwards HM, Sort R, Vilandt J, Gogenur I. Translation and validation of the Danish version of the postoperative quality of recovery score QoR-15. Acta Anaesthesiol Scand. 2015 Aug;59(7):912-20. doi: 10.1111/aas.12525. Epub 2015 Apr 13. PMID 25867135
- [Result] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Result] Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA; AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest. 2001 Feb;119(2):590-602. doi: 10.1378/chest.119.2.590. PMID 11171742
- [Result] Akamine T, Kometani T, Hashinokuchi A, Akamine S, Shikada Y, Wataya H. Interpleural distance predicts persistent air leak after initial primary spontaneous pneumothorax. J Thorac Dis. 2020 May;12(5):2228-2235. doi: 10.21037/jtd.2020.04.48. PMID 32642128
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Hansen HJ, Petersen RH. Video-assisted thoracoscopic lobectomy using a standardized three-port anterior approach - The Copenhagen experience. Ann Cardiothorac Surg. 2012 May;1(1):70-6. doi: 10.3978/j.issn.2225-319X.2012.04.15. No abstract available. PMID 23977470
- [Result] Zhou Q. [Recommendations for the conduct, reporting, editing and publication of scholarly work in medical journals]. Zhonghua Gan Zang Bing Za Zhi. 2014 Oct;22(10):781-91. No abstract available. Chinese. PMID 25558501
- [Derived] Holbek BL, Huang L, Christensen TD, Bendixen M, Hansen HJ, Kehlet H, Petersen RH. Efficacy of avoiding chest drains after video-assisted thoracoscopic surgery wedge resection: protocol for a randomised controlled trial. BMJ Open. 2024 Feb 20;14(2):e080573. doi: 10.1136/bmjopen-2023-080573. PMID 38382951